CLINICAL TRIAL: NCT02059447
Title: A Comparison of the Benefits of Mindfulness Based Cognitive Therapy, Relaxation Therapy and a Waiting List Control in the Management of Distress in Chronic Tinnitus Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College London Hospitals (Other)
Collaborators: University College, London (Other); British Tinnitus Association (Other)
Responsible Party: Principal Investigator, Dr Laurence McKenna, Clinical psychologist, University College London Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tinnitus MBCT
Record Dates: First submitted 2014-01-24; First posted 2014-02-11 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Tinnitus
Keywords: Controlled trial; Active control; Waiting, non treatment, period; Mindfulness Based Cognitive Therapy; Relaxation Therapy
MeSH Terms: conditions — Tinnitus | interventions — Mindfulness-Based Cognitive Therapy; Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness Based Cognitive Therapy (Experimental): An 8 week course of Mindfulness Based Cognitive therapy
  Interventions: Other: No treatment waiting period; Behavioral: Mindfulness Based Cognitive Therapy
- Relaxation Therapy (Active Comparator): An 8 week course of Relaxation Therapy.
  Interventions: Other: No treatment waiting period; Behavioral: Relaxation Therapy

INTERVENTIONS:
Other: No treatment waiting period — All subjects undergo a no treatment waiting period before being randomly allocated to either Mindfulness Based Cognitive Therapy or Relaxation Therapy
Behavioral: Mindfulness Based Cognitive Therapy
  Arms: Mindfulness Based Cognitive Therapy
Behavioral: Relaxation Therapy
  Arms: Relaxation Therapy

SUMMARY:
The principal hypotheses to be tested is that Mindfulness Based Cognitive Therapy (MBCT) reduces the distressing impact of tinnitus to a significantly greater extent than a waiting list control or relaxation therapy.

This study is a mixed design, with two groups assessed at a number of time points. The primary outcome measure will be that of tinnitus distress, and secondary outcomes will be taken of psychological distress and tinnitus loudness.

The outcome measures will be measured first at 8 weeks pre-treatment. All subjects then wait for 8 weeks before being randomly allocated to either an 8 week course of Mindfulness-Based Cognitive Therapy (MBCT) (Group 1) or an 8 week course of Relaxation Therapy (RT) (Group 2). All participants will be assessed at two main time-points (pre and post-treatment). The outcome measures will be repeated at 1 and 6 month follow-up points.

DETAILED DESCRIPTION:
Experimental design and methods (including statistical analysis)

Participant recruitment:

Potential participants who meet the eligibility criteria will be identified from among patients referred to the adult clinical psychology service within the department of Adult Audiology at the Royal National Throat Nose & Ear Hospital. These patients will be approached and invited to discuss participation in the project. The potential participants will be given full information about the study and invited to consider whether they wish to participate.

Design

This study an independent groups, repeated measures design. Two groups will be assessed at different time points. Group 1 will receive 8 weeks of Mindfulness-Based Cognitive Therapy (MBCT) and Group 2 will receive 8 weeks of Relaxation Training (RT; an active control). All participants will be assessed at five main time-points:

* 8 weeks pre-treatment,
* The start of treatment
* The end of treatment
* 1 month follow-up
* 6 month follow-up

The primary outcome measure will be that of tinnitus complaint, and secondary outcome measures will be taken of psychological distress and tinnitus loudness, tinnitus acceptance and everyday mindfulness.

Measures:

A number of Questionnaire measures and a Visual Analogue Scale will be used to assess tinnitus complaint, psychological well-being and mindfulness.

Participants are evaluated on all measures at initial assessment (8 weeks pre-treatment), at treatment commencement, at end of treatment and at 1and 6 month follow-up.

Statistical Analyses

The primary outcome will be the change in tinnitus complaint as measured by the Tinnitus Questionnaire from pre-treatment to post-treatment. This will be assessed by using t-tests.

Further statistical exploration will use t-tests to assess change from initial assessment to end of the 8-week waiting period, and to assess change or maintenance of change from the end of treatment to the 1and 6 month follow-up points. The same type of analysis will be done on the measures of psychological well-being.

To assess for differences in outcome between the MBCT and RT groups, a series of repeated-measures (2x2) (Group 1 - Group 2 x pre-treatment - post-treatment) ANOVAS will be carried out. This will allow for the assessment of between group effects and any interaction effects between group and time.

A number of correlations will also be performed to assess for relationships between psychological distress pre-treatment and tinnitus outcome within each group. Correlation will also be performed to assess for relationships between changes in tinnitus complaint and tinnitus acceptance and everyday mindfulness. They will also be performed to assess for relationships between changes in psychological distress and everyday mindfulness.

Chi-square analyses will be carried out on the measures of tinnitus complaint and CORE-OM score pre- and post-treatment to assess for the numbers of patients within each group who demonstrate clinically significant change. A clinically significant change in tinnitus complaint is defined as change of at least 10 points reduction on the TQ. A clinically significant change in psychological well-being is defined as a reduction of at least 0.5 on the total mean CORE-OM score.

Correlations will be performed to assess for possible associations between patient characteristics, attendance, amount of home practice and various outcomes. Weekly measures of mindfulness will be used to explore the temporal sequence of change.

Methodology:

All participants will be assessed using all of the measures described above over a 2 week period. They will then be randomly assigned to one of two groups: Group 1 will be treated using an 8 week course of Mindfulness-Based Cognitive Therapy (MBCT). Group 2 will be treated using an 8 week course of Relaxation Training (RT).This randomization will be carried out by a member of staff at the Ear Institute, who is independent from the clinical part of the trial. He will use a computer programme to complete randomization.

After assessment, patients enter a 'waiting' stage of the trial, during which they receive no intervention for eight weeks. Four weeks into the waiting time, all patients will be sent a letter to confirm the dates and times at which their specific group will take place. On the eighth week, participants will attend the first group session. At this point, prior to commencement of the group, they will complete all of the measures described above for a second time.

All participants will then attend 8 consecutive weeks of group treatment. Throughout this treatment period, at the end of each session, participants will complete two brief measures (the MAAS the TAQ). This is important as it will allow for the temporal sequence of change to be assessed, offering an opportunity to explore the potential mediation effect of mindfulness. At the end of the eighth week, they will again be asked to complete all of the measures for a third time.

All participants will then be invited to attend two further sessions - at 1 and 6 months after treatment completion. At the start of these sessions all participants will be asked to complete all of the measures described above for a fourth and fifth time. These sessions will also provide ongoing support to the participants as they will provide an opportunity to discuss how they are after the groups have finished.

Thus MBCT will be compared to an active control condition (RT) and a passive control condition (wait list control), and RT will also be compared to the passive wait-list control condition.

ELIGIBILITY:
Inclusion Criteria:

1. Only patients with chronic tinnitus (i.e. have had tinnitus for six months or more) will be included
2. Only patients who show at least a minimum level of distress (defined by a cut off score on the CORE measure of psychological well-being).
3. Only patients whose hearing permits them to take part in group discussions in a quiet room will be included.
4. Only patients with sufficient understanding of English to take part in group discussions and complete questionnaires will be included.

Exclusion Criteria:

1. Patients who are subject to ongoing medical investigations will be excluded. Patients who are alcohol or drug dependent will be excluded Patients who are suffering with psychosis or who are actively suicidal will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in Tinnitus Questionnaire score over time | 8 weeks pre treatment; start of treatment; end of treatment; 1 month post treatment; 6 months post treatment

SECONDARY OUTCOMES:
Change in Clinical Outcomes in Routine Evaluation (Outcome measure) score over time | 8 weeks pre treatment; start of treatment; end of treatment; 1 month post treatment; 6 months post treatment

OTHER OUTCOMES:
Change in Tinnitus Functional Index score over time | 8 weeks pre treatment; start of treatment, end of treatment, 1 month post treatment; 6 months post treatment
Change in Mindful Attention Awareness Scale score over time | 8 weeks pre treatment; start of treatment; end of treatment, 1 month post treatment; 6 months post treatment
Change in Tinnitus Acceptance Questionnaire score over time | 8 weeks pre treatment; start of treatment; end of treatment; 1 month post treatment; 6 months post treatment
Change in Visual Analogue Scalescore over time | 8 weeks pre treatment; start of treatment; end of treatment; 1 month post treatment; 6 months post treatment
Change in Hospital Anxiety and Depression Scale score over time | 8 weeks pre treatment; start of treatment; end of treatment; 1 month post treatment; 6 months post treatment
Change in Tinnitus Fear Avoidance Scale over time | 8 weeks pre treatment, start of treatment, end of treatment, 1 month post treatment; 6 months post treatment
Change in Tinnitus Catastrophy Scale score over time | 8 weeks pre treatment, start of treatment, end of treatment, 1 month post treatment; 6 months post treatment
Change in Work & Social Adjustments Scale score over time | 8 weeks pre treatment, start of treatment, end of treatment, 1 month post treatment; 6 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Laurence McKenna, PhD, Principal Investigator — Royal National Throat Nose & Ear Hospital, University College London Hospitals
Locations (1):
- Royal National Throat Nose & Ear Hospital, University College London Hospitals, London, England, United Kingdom